CLINICAL TRIAL: NCT02425878
Title: Uterine Fibroids: Impact of Ulipristal Acetate 10 mg on ART Results
Brief Title: Ulipristal Acetate 10 mg and Asisted Reproduction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of availibility of eligible subjects
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1311-BCN-138-DG
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Intramural Fibroids; Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Ulipristal Acetate 10 mg, Oral administration. Dose: 10 mg per day, single dose, duration 12 weeks
  Interventions: Drug: Ulipristal Acetate
- Control (Placebo Comparator): Placebo, 10 mg, Oral administration. Dose: 10 mg per day, single dose, duration 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulipristal Acetate
  Arms: Experimental
Drug: Placebo
  Arms: Control

SUMMARY:
Demonstrate an 15% increase in the rate of clinical pregnancy in women with inoperable intramural fibroids not distorting the uterine cavity within a program OVD, after administration of uPA in a dose of 10 mg orally daily for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

Patients> 18 and <50 years Patients who undergo a first / second cycle OVD Patients who present within 1-3 intramural myomas> 2 cm and <5 cm that do not distort the cavity, Type 3 and 4 of the FIGO classification (Figure 1). Miomas inoperable for medical judgment or patient desire, you want to avoid the post-surgical time waiting 6 months / 1 year before you can submit to TRA Patients who have undergone previous myomectomy who prefer to avoid having surgery

Exclusion Criteria:

History of endometrial changes in patients (hyperplasia) Presence of other endometrial pathologies: polyps, scars of previous cesarean complicated adenomyosis foci, suspected adhesions Simultaneous participation in another clinical study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
increase in the rate of clinical pregnancy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Galliano, MDPhD, Principal Investigator — Instituto Valenciano de Infertilidad, IVI VALENCIA
Locations (1):
- IVI Valencia, Valencia, Spain